CLINICAL TRIAL: NCT03265639
Title: Prebiotics in Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Ramezani (Other)
Responsible Party: Sponsor-Investigator, Ali Ramezani, Assistant Research Professor, George Washington University
Organization: George Washington University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 091440
Record Dates: First submitted 2017-02-17; First posted 2017-08-29 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: End Stage Renal Disease; Gut Microbiome Dysbiosis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-treatment (No Intervention): This arm is the 8-week observation period before the p-inulin treatment phase.
- Intervention (Experimental): This arm is the 8 week p-inulin treatment phase (8 grams twice daily, oral).
  Interventions: Dietary Supplement: P-inulin
- Post-treatment (No Intervention): This arm is the 8-week observation period after the p-inulin treatment phase.

INTERVENTIONS:
Dietary Supplement: P-inulin
  Arms: Intervention

SUMMARY:
The Prebiotics in Peritoneal Dialysis trial is a non-randomized, open-label, crossover study of p-inulin for patients with end-stage renal disease treated with peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis therapy for end-stage renal disease
* ≥30 days since dialysis initiation
* Ability to provide informed consent

Exclusion Criteria:

* Use of pre- or pro-biotics during the past 2 months
* Consumption of pro-biotic yogurt during the past 2 weeks
* Use of antibiotics within the past 2 months
* Presence of chronic infection
* Chronic gastrointestinal condition other than constipation
* Cirrhosis or chronic active hepatitis
* Stomach/intestinal resection
* PD access problems
* Anticipated kidney transplant or transfer to another dialysis unit within 9 months
* Expected survival < 9 months
* Pregnancy, anticipated pregnancy, or breastfeeding
* Incarceration
* Participation in another intervention study
* Severe anemia defined as hemoglobin <9.0 g/dl

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change within-patient in the metabolomic profile and targeted metabolites / inflammatory markers during the no treatment phases and the p-inulin treatment phase. | 24 weeks
  Metabolomic Profile: the relative abundance of metabolites, determined by liquid chromatography-mass spectrometry (LC-MS), will be quantified under each condition and compared between groups.

SECONDARY OUTCOMES:
Within-patient change in the metabolomic profile and targeted metabolites / inflammatory markers after p-inulin treatment compared with pre-treatment. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Metabolomic Profile: the relative abundance of metabolites, determined by liquid chromatography-mass spectrometry (LC-MS), will be quantified under each condition and compared between groups.
Within-patient variability in the bacterial composition of the stool during the no treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified.
Within-patient variability in the bacterial composition of the stool during the p-inulin treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified.
Within-patient change in the bacterial composition of the stool after p-inulin treatment compared with pre-treatment | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified.
Within-cohort variability in the metabolomic profile and targeted metabolites / inflammatory markers during the no treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Metabolomic Profile: the relative abundance of metabolites, determined by liquid chromatography-mass spectrometry (LC-MS), will be quantified under each condition and compared between groups.
Within-cohort variability in the bacterial composition during the no treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified under each condition and compared between groups.
Within-cohort variability in the metabolomics profile and targeted metabolites/inflammatory markers during the p-inulin treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Metabolomic Profile: the relative abundance of metabolites, determined by liquid chromatography-mass spectrometry (LC-MS), will be quantified under each condition and compared between groups.
Within-cohort variability in the bacterial composition during the p-inulin treatment phase. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified under each condition and compared between groups.
Within-cohort change in the metabolomic profile and targeted metabolites/inflammatory markers after p-inulin treatment compared with pre-treatment | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Metabolomic Profile: the relative abundance of metabolites, determined by liquid chromatography-mass spectrometry (LC-MS), will be quantified under each condition and compared between groups.
Within-cohort change in the bacterial composition after p-inulin treatment compared with pre-treatment. | 24 weeks (8 week period of observation, 8 week period of treatment, 8 week period of observation)
  Bacterial Composition: the relative abundance of bacterial taxa, as determined by 16S rRNA gene sequencing, will be quantified under each condition and compared between groups.

OTHER OUTCOMES:
Change in Score of the Gastrointestinal Symptom Rating Scale (GSRS) | 24 weeks
  Gastrointestinal symptoms as measured by the Gastrointestinal Symptom Rating Scale (GSRS)
Number of Participants Who Discontinue Use of p-inulin | 8 week period of treatment
Number of Participants Who Reduce the Dose of p-inulin | 8 week period of treatment
Number of Adverse Events | 24 weeks
Enrollment Refusal Rate | 2 years
Proportion of completed stool sample collections | 24 weeks
Proportion of completed blood sample collections | 24 weeks
Adherence rate to p-inulin | 8 weeks
  Assessed by sachet counts
Rate of Study Withdrawal | 24 weeks
  Number of subjects who withdrew during each phase

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Raj, MD, Principal Investigator — The George Washington University
Locations (2):
- United States (2):
  - DaVita Georgetown Home Training Unit, Washington D.C., District of Columbia
  - DaVita K Street, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No